CLINICAL TRIAL: NCT04003753
Title: Randomized Controlled Trial on the Efficacy of a Virtual Reality Paradigm to Reduce Fear of Heights in a Clinical and Subclinical Population With Fear of Heights
Brief Title: Efficacy of a VR Paradigm to Reduce Fear of Heights in a Clinical and Subclinical Population With Fear of Heights
Acronym: VRAP-Basel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Prof Dr. med., University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-01504
Record Dates: First submitted 2019-06-24; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Fear of Heights
MeSH Terms: conditions — Acrophobia

STUDY DESIGN:
Intervention Model Description: randomized controlled single-blind study design
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly (matched by clinical relevance of fear of heights and sex) allocated to treatment groups (experimental group, control group). The experimenter evaluating the primary outcome will be blinded (unaware of group assignment of participants, single-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure (Experimental): Study phase 1: The experimental intervention in the experimental group consists of three 20-minutes VR exposures (total duration in VR: 60 minutes).
  Study phase 2: The experimental intervention in the experimental group consists of six 30-minutes VR exposures as home training (total duration in VR: 3 hours) within two weeks.
  Interventions: Other: VR App
- Control (No Intervention): Study phase 1: The control group will not receive any active treatment. Instead they will use an App to make virtual tours (three times 20 minutes, total duration in VR: 60 minutes).
  Study phase 2: The control group will not receive any active treatment (untreated comparison group).

INTERVENTIONS:
Other: VR App — Participants will be exposed in three different virtual height scenarios (rural mountain, urban town, cloudy weather). At the beginning of each exposure session participants will be standing on a virtual platform at ground level (level 0). From level 0 they will proceed to further levels according to a predefined exposure scheme based on SUDS ratings (scale 0=no fear to 10=extreme fear). Participants will have to stay at each level until their SUDS are 3 or below for two times consecutively (assessment via gaze selection). In each scenario there will be 15 different height levels available (corresponding to a range of heights between 1-75m). Each exposure session will be terminated by a time limit of 20 minutes (study phase 1) or 30 minutes (study phase 2) irrespective of achieved level.
  Arms: Exposure

SUMMARY:
Investigation of the effectiveness and acceptability and usability of a VR height exposure App in individuals with fear of heights.

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled between subject trial. The study consists of two study phases. In study phase 1 the experimental group takes part in three VR exposure sessions (duration 20min each), whereas the control group takes part in three virtual tours (duration 20min each). All VR sessions and assessments of outcomes will be conducted on one study day for each participant.

In study phase 2 the experimental group will participate in a home training, spanning over two weeks (6x30-minutes sessions), whereas the control group will not receive any treatment (untreated comparison group). Assessment of outcomes will be conducted 3-5 weeks after completion of home trainings.

Group 1 (experimental group) consists of individuals with clinical and subclinical fear of heights, that will receive a three-session VR exposure (study phase 1) and take part in a 2-week treatment period with the same VR scenarios (study phase 2). Group 2 (control group) consists of individuals with clinical and subclinical fear of heights that will not receive any active treatment, but will participate in fear-unrelated tasks in study phase 1 or receive no treatment at all (study phase 2).

This design allows a direct comparison and therefore an estimation of the effectiveness of the VR exposure therapy. Before and after the virtual exposure/tours participants will undergo an in vivo BAT to assess the effects of the VR exposure therapy.

80 participants between 18 and 60 years with clinical or subclinical fear of heights will take part in the study. Two to three months after having finished study phase 1 the participants will be contacted again and asked to take part in study phase 2. All participants undergo a third in vivo BAT during study phase 2. The BAT will take place 3-5 weeks after completion of the home training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical fear of heights (DSM-V) or subclinical fear of heights (fulfilment of DSM-C criteria A-E and G, but not F: distress/impairment)
* Physically healthy
* Aged between 18-60
* Fluent in German

Exclusion Criteria:

* Depression (BDI-II > 8)
* Suicidal ideation (BDI-II item 9 > 0)
* Concurrent psychotherapy or pharmacotherapy
* Previous therapy for height phobia
* Parallel participation in another study
* Pregnancy (will be excluded with a pregnancy test during screening)
* Chronic medication intake (except oral contraceptives)
* Alcohol and medication intake before visit (less than 12 h)
* Cannabis or other psychoactive substances (including benzodiazepines) intake before visit (less than 5 days)
* Sleep-inducing drugs (incl. antihistamines) intake before visit (less than five days)
* Restricted 3D sight

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Performance Behavioural Avoidance Test (BAT) in vivo | study phase 1: on study day within 1h after VR exposure, study phase 2: 3-5 weeks after completion of home training
  Change in BAT performance after VR exposure from baseline (before VR exposure). During the BAT participants will be requested to climb up to the Uetliberg Tower while continuously looking to the ground level. Participants will be asked to only proceed as far as their anxiety allows them. On each of the 14 platforms participants will be asked to lean on a predefined area of the railing (and touch it with their upper body) and to look down to the ground for 10 seconds, if their fear allows them to do so. The BAT will be terminated as soon as the participant indicates feeling uncomfortable to proceed (adapted from Emmelkamp, 2002 and Coelho, 2006) or the 10 minutes period, given to them to perform the complete task, runs out.

SECONDARY OUTCOMES:
Acrophobia Questionnaire (AQ) | study phase 1: on study day within 1h after VR exposure, study phase 2: 3-5 weeks after completion of home training
  Change in AQ after VR exposure from baseline (before VR exposure).This questionnaire describes twenty situations that can cause fear of heights (e.g., driving over a bridge, walking over a sidewalk grating, or sitting on an airplane) and asks for anxiety ratings on a 7-point Likert-type scale (0 = not at all afraid to 6 = very afraid, range 0-120, α = 0.80) (Cohen, 1977).
Attitudes Towards Heights Questionnaire (ATHQ) | study phase 1: on study day within 1h after VR exposure, study phase 2: 3-5 weeks after completion of home training
  Change in ATHQ after VR exposure from baseline (before VR exposure).The ATHQ consists of six questions assessing participants' attitudes towards heights situations (e.g., "I think heights are … good - bad, secure - insecure"). Patients evaluate their attitudes towards heights by twelve adjectives on an 11-point scale ranging from a positive (0) to a negative (10) adjective (range 0-60; α = 0.81).
Anxiety Expectancy Scale (AES) | study phase 1: on study day within 1h after VR exposure, study phase 2: 3-5 weeks after completion of home training
  Change in AES after VR exposure from baseline (before VR exposure). The AES assesses anxiety symptoms in a height situation. The AES consists of ten items describing anxiety symptoms (e.g., "you could feel dizzy"). Participants rate the likelihood of experiencing these symptoms while being in a height situation on a five-point scale (range 10-50) (Gursky & Reiss, 1987).
Danger Expectancy Scale (DES) | study phase 1: on study day within 1h after VR exposure, study phase 2: 3-5 weeks after completion of home training
  The DES assesses dysfunctional cognitions. The DES consists of five items. Participants rate the likelihood that each of the listed harmful events (e.g., "you might slip and fall over the guard rail on the observation deck") will pass through their minds while being in a height situation on a five-point scale (not likely at all (1), probably not (2) maybe (3), quite likely (4), or definitely (5), range 5-25) (Gursky & Reiss, 1987).

OTHER OUTCOMES:
VR exposure app acceptability and usability scale | study phase 1: on study day within 1h after VR exposure, study phase 2: 3-5 weeks after completion of home training
  The VR exposure app acceptability and usability scale consists of 10 items (study phase 1)/11 items (study phase 2) that assess the overall acceptability and usability (e.g. design, functionality) of the VR app. The items were solely composed for our study purposes. The first 9 items will be assessed through a 11-point scale, item 10 and 11 have an open answer format. Higher scores indicate higher acceptability and usability.
Igroup Presence Questionnaire (IPQ) | study phase 1: on study day directly (within 1h) after VR exposure
  The IPQ assess participants' presence while being in VR. The IPQ consists of 14 items with a 7-point scale (0-6) that concern the participants' sense of being in the virtual environment, for example, the extent to which virtual reality was "real" to them, whether they thought of the virtual environment more as images they saw or more as a situation they were in, how much attention they paid to the real world, and the extent to which they focused on the virtual task. The IPQ consists of three subscales: Spatial Presence (range 0-30), Involvement (range 0-24), Realness (range 0-12), higher scores indicate stronger presence (Schubert, 2003).
Subjective Units of Distress Scale (SUDS) | on study day during VR exposure
  Participants in the experimental group will be prompted to give their SUDS during the VR heights exposure sessions at predefined time points (first rating on each level after 10 seconds, then every 30 seconds until allowed to enter the next level. Then again first rating after 10 seconds, then every 30 seconds until allowed to enter the next level and so on (scale 0=no fear to 10=extreme fear).
Simulator Sickness Questionnaire (SSQ) | study phase 1: on study day directly (within 1h) after VR exposure
  Assessment of potential side effects of VR immersion. Possible symptoms (e.g. headache, nausea) will be assessed directly before (baseline) and after the VR exposure on a scale between 0-3. The change from baseline will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof., Principal Investigator — University of Basel
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland